CLINICAL TRIAL: NCT05996822
Title: Evaluation of Diabetic or Uveitic Macular Edema After Injection of a Fluocinolone Acetonide (AcF) Implant 1 Month After the Last Dexamethasone (DXM) Implant: Evaluation at 3 Years
Brief Title: Evaluation of Macular Edema After AcF Implant's Injection, 1 Month After the Last DXM Implant
Acronym: ILUV1MOIS2
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_JBD_002
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — A1CF protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AcF injection: Patient having received an AcF injection 1 month after a DXM injection for the treatment of Diabetic Macular Edema or Uveitic Macular Edema
  Interventions: Drug: ACF injection

INTERVENTIONS:
Drug: ACF injection — AcF injection 1 month after a DXM injection

SUMMARY:
Patients with diabetic macular edema (DME) or uveitis-related macular edema who have failed first-line therapy such as anti-VEGF, laser treatments, or dexamethasone implants (DXM) are candidates for treatment with an intravitreal injection of a fluocinolone acetonide (AcF) implant. AcF is unique in that it delivers intravitreal corticosteroids for 2 to 3 years, whereas DXM only releases them for 3 to 6 months. After 6 months for AcF and 1 month for DXM, full therapeutic efficacy is attained.

AcF's safety and efficacy have now been confirmed in the FAME originator studies as well as other phase IV investigations. However, in the FAME princeps trials and numerous phase IV trials where patients got AcF more than 6 months after DXM, up to 40% of patients required laser, anti-VEGF, and/or DXM retreatment within the AcF active period. This high rate could be attributed to AcF's 6-month delay in reaching full efficacy.

This is why the investigators intended to replicate the previous Iluvi1-month research, which shown that injecting DXM at 1 month preserved visual acuity and central retinal thickness for the first 6 months without increasing intraocular pressure significantly. The study, however, was unable to determine the long-term impact on the rate of relapses requiring additional therapy as well as tolerance with the development of long-term cortisone-induced glaucoma.

In light of this, the investigators should like to gather new data for a 3-year follow-up after AcF injection, including measurements of optic nerve fibre thickness (OCT RNFL). This is an essential safety data point because it assesses the long-term effects of ocular hypertension, which is a well-known side effect of intravitreal corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Patient (Male, Female)°≥ 18 years old
* Having received an AcF injection 1 month after a DXM injection
* For diabetic macular edema or uveitic macular edema

Exclusion Criteria:

* Patient's refusal to allow his or her medical data to be used for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants recruited in the study extension will be the same as those in the initial ILUV1MOIS study.
  The investigators will present the study extension to the patients at their scheduled routine care visits.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Efficiency (ETDRS) | 1 month after AcF injection
  change in visual acuity by ETDRS between baseline(before AcF injection) and 1 month after

SECONDARY OUTCOMES:
Efficiency (OCT) | 1 month after AcF injection
  change in macular thickness by OCT between baseline(before AcF injection) and 1 month after
safety (AE) | 1 month after AcF injection
  Report of the adverse events during 1 month after ACF injection

CONTACTS AND LOCATIONS:
Locations (1):
- Jean-Baptiste Ducloyer, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided